CLINICAL TRIAL: NCT03171129
Title: Adaptive Dynamic Inspiratory Nasal Apparatus (ADINA): Comparison to High Flow Nasal Cannula (HFNC)
Brief Title: ADINA vs. High Flow Nasal Cannula Comparison Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5160055
Record Dates: First submitted 2017-05-25; First posted 2017-05-31 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Distress Neonatal
Keywords: Respiratory Distress; Nasal CPAP; high flow nasal canula
MeSH Terms: conditions — Hyaline Membrane Disease; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- High flow nasal cannula system w/ ADINA (Experimental): The intervention is the insertion of the the ADINA device into the high flow nasal cannula system. ADINA will be placed according to weight class recommendations to increase the positive end expiratory pressure (PEEP). ADINA is actually a combination of the Neotech RAM Cannula and a clear Regulator/Pop off valve.
  Interventions: Device: Adaptive Dynamic Inspiratory Nasal Apparatus
- high flow nasal cannula system (Active Comparator): High flow nasal cannula will deliver oxygen at 2-4 lpm of flow. High flow cannula are used to provide the control interface.
  Interventions: Device: High flow Nasal Canula

INTERVENTIONS:
Device: Adaptive Dynamic Inspiratory Nasal Apparatus — Oxygen will be administered via ADINA
  Other Names: ADINA
  Arms: High flow nasal cannula system w/ ADINA
Device: High flow Nasal Canula — Oxygen will be administered via nasal canula
  Arms: high flow nasal cannula system

SUMMARY:
This study is to evaluate the feasibility of using a pressure limited nasal cannula system instead of a high flow nasal cannula system in the management of premature babies with respiratory distress.

DETAILED DESCRIPTION:
NCPAP has been used increasingly to manage respiratory distress in newborns as well as apnea of prematurity. Humidified high flow nasal cannula devices (flows 1-8 lpm) have also been used in neonatal intensive care units.

This study is to evaluate the feasibility of using a pressure limited nasal cannula system instead of a high flow nasal cannula system in the management of premature babies with respiratory distress.

ELIGIBILITY:
Inclusion Criteria:

* Neonates admitted to NICU
* Weights of 400-500 grams
* Requiring oxygen greater than 30%
* No evidence of focal lobar consolidation in lung fields

Exclusion Criteria:

* Intolerance to procedure
* gelatinous skin
* known allergy to adhesive material
* interference with therapy
* profound sepsis
* pneumonia
* unmanaged apnea/bradycardia
* known or suspect complex congenital heart disease
* severe cleft lip or palate
* suspect or proven lethal congenital anomaly
* intolerance to the interface used in the devices
* inability to secure an appropriate fit of the patient nasal interface
* considered non-viable or of uncertain viability
* parental refusal.

Ages: 23 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Duration of Oxygen Use | From time of randomization until time of discharge from the Neonatal Intensive Care Unit (NICU) up to 100 days.
  The length of time the patient is on oxygen will be measured in hours.

SECONDARY OUTCOMES:
Oxygen Concentration | From time of randomization until time of discharge from NICU up to 100 days.
  ADINA will provide a concentration of oxygen between 1.5 and 4 liters which is equivalent to that provided by the conventional nasal cannula. This will be measured every twelve hours by NICU staff.
Number of Participants with treatment-related pneumothorax | From time of randomization until time of discharge from NICU up to 100 days.
  Participants will be monitored for pneumothorax occurrence while on ADINA and/or high flow nasal cannula. The incidence of pneumothorax occurrence in each Arm will be collected for comparison.
Number of Participants with Excoriation at Nasal Site | From time of randomization until time of discharge from NICU up to 100 days.
  Participants will be monitored for excoriation at the nasal site while on ADINA and/or high flow nasal cannula. The incidence of excoriation at the nasal site in each Arm will be collected for comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell R Goldstein, MD, Principal Investigator — Loma Linda University Health
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gregory GA, Kitterman JA, Phibbs RH, Tooley WH, Hamilton WK. Treatment of the idiopathic respiratory-distress syndrome with continuous positive airway pressure. N Engl J Med. 1971 Jun 17;284(24):1333-40. doi: 10.1056/NEJM197106172842401. No abstract available. PMID 4930602
- [Background] Dutta S. High-flow nasal cannula versus nasal continuous positive airway pressure in the management of apnea of prematurity. Pediatrics. 2002 Apr;109(4):718-9; author reply 718-9. doi: 10.1542/peds.109.4.718. No abstract available. PMID 11927724
- [Background] Campbell DM, Shah PS, Shah V, Kelly EN. Nasal continuous positive airway pressure from high flow cannula versus Infant Flow for Preterm infants. J Perinatol. 2006 Sep;26(9):546-9. doi: 10.1038/sj.jp.7211561. Epub 2006 Jul 13. PMID 16837929
- [Background] Kubicka ZJ, Limauro J, Darnall RA. Heated, humidified high-flow nasal cannula therapy: yet another way to deliver continuous positive airway pressure? Pediatrics. 2008 Jan;121(1):82-8. doi: 10.1542/peds.2007-0957. PMID 18166560
- [Background] Woodhead DD, Lambert DK, Clark JM, Christensen RD. Comparing two methods of delivering high-flow gas therapy by nasal cannula following endotracheal extubation: a prospective, randomized, masked, crossover trial. J Perinatol. 2006 Aug;26(8):481-5. doi: 10.1038/sj.jp.7211543. Epub 2006 May 25. PMID 16724119
- [Background] Shoemaker MT, Pierce MR, Yoder BA, DiGeronimo RJ. High flow nasal cannula versus nasal CPAP for neonatal respiratory disease: a retrospective study. J Perinatol. 2007 Feb;27(2):85-91. doi: 10.1038/sj.jp.7211647. PMID 17262040
- [Background] Sreenan C, Lemke RP, Hudson-Mason A, Osiovich H. High-flow nasal cannulae in the management of apnea of prematurity: a comparison with conventional nasal continuous positive airway pressure. Pediatrics. 2001 May;107(5):1081-3. doi: 10.1542/peds.107.5.1081. PMID 11331690
- [Background] Centers for Disease Control and Prevention (CDC). Update: Ralstonia species associated with Vapotherm oxygen delivery devices--United States, 2005. MMWR Morb Mortal Wkly Rep. 2005 Nov 4;54(43):1104-5. PMID 16267498
- [Background] Centers for Disease Control and Prevention (CDC). Ralstonia associated with Vapotherm oxygen delivery device--United States, 2005. MMWR Morb Mortal Wkly Rep. 2005 Oct 21;54(41):1052-3. PMID 16237377